CLINICAL TRIAL: NCT07323173
Title: A Phase I, Double-Blind, Randomized, Placebo-Controlled, Dose-Escalation Study of Single Subcutaneous Injections of LBL-047 in Healthy Adults and Patients With Systemic Lupus Erythematosus
Brief Title: A Phase I Study to Assess LBL-047 in Healthy Adults and Patients With Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Collaborators: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBL-047-CN001
Record Dates: First submitted 2025-11-29; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBL-047 for Injection (Experimental): LBL-047 for Injection,Single subcutaneous injection.
  Interventions: Drug: LBL-047 for Injection
- LBL-047 placebo for injection (Active Comparator): LBL-047 placebo for injection,Single subcutaneous injection.
  Interventions: Drug: LBL-047 placebo for injection

INTERVENTIONS:
Drug: LBL-047 for Injection — Single subcutaneous injection
  Other Names: LBL-047
  Arms: LBL-047 for Injection
Drug: LBL-047 placebo for injection — Single subcutaneous injection
  Other Names: LBL-047 placebo
  Arms: LBL-047 placebo for injection

SUMMARY:
A Phase I, Double-Blind, Randomized, Placebo-Controlled, Dose-Escalation Study of Single Subcutaneous Injections of LBL-047 in Healthy Adults and Patients with systemic lupus erythematosus.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled Phase I study to evaluate the safety, tolerability, PK, PD and immunogenicity of a single subcutaneous injection of LBL-047 in healthy adults and patients with systemic lupus erythematosus,the preliminary clinical efficacy of LBL-047 will also be evaluated in patients with systemic lupus erythematosus.

The study is divided into two parts.

Part A:Conduct studies in healthy adults.Part A is planned to be set up with 7 escalating dose groups.Participants were randomized to receive a single subcutaneous injection of LBL-047 or placebo.Dose escalation will be decided by the Safety Monitoring Committee (SMC).

Part B:Study in adult patients with systemic lupus erythematosus.Part B will be initiated at the dose levels that were confirmed to be safe and tolerable in Part A.Part B is planned to enroll patients with mild to moderate systemic lupus erythematosus and receive a single subcutaneous injection of LBL-047.

This study is expected to enroll 76 participants (with possible addition of 36 participants).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign and date the informed consent form (ICF) and be willing and able to comply with the scheduled visits, treatment plan, laboratory test, and other study procedures.
2. Age ≥ 18 and ≤ 60 years at the time of signing the ICF.
3. Part A:Determined by the investigator to be in good health at the time of signing the ICF.
4. Part B:Mild to moderate systemic lupus erythematosus: SLEDAI-2K score ≥4 and ≤ 10 at screening.
5. Females of childbearing potential are willing to use highly effective contraception during the study and for 6 months after administration of the study drug and to avoid egg donation.Women of non-childbearing potential include: those with documented surgical sterilization or documented menopause.
6. Male of childbearing potential are willing to use highly effective contraception during the study and for 6 months after study drug administration and to avoid sperm donation.Men without fertility potential include those with: A semen sample investigation that confirms azoospermia, definitive evidence of infertility, or a history of vasoligation.For the purpose of this study, men with a "low sperm count" (or "subfertility") are not considered infertile.

Exclusion Criteria:

1. Part A:Symptoms or history of any significant disease, including but not limited to cardiovascular, hepatic, renal or any other disease that may interfere with the study results.
2. Part A:Abnormalities with clinical significance were indicated by vital signs, physical examination, laboratory test, 12-lead electrocardiogram (ECG), chest X-ray, and abdominal ultrasound.
3. Part B:History of organ transplant or hematopoietic stem cell/bone marrow transplant.
4. Part B:currently receiving treatment for any chronic infection (such as pneumocystosis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteriosis).
5. Major surgery (as judged by the investigator) within 90 days prior to dosing, or surgery scheduled during the study.
6. At screening, women of childbearing potential were positive for pregnancy.follicle stimulating hormone (FSH) did not reach postmenopausal level in postmenopausal women (defined as amenorrhoea ≥ 12 months before screening).
7. Large tattoo, scar or other condition that may interfere with assessment at the injection site.
8. unable to tolerate venipuncture, difficulty in blood collection or has a history of needle/blood phobic disorder.
9. The investigator determines that there are other conditions unsuitable for participation in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2027-12-16 (Estimated); Study Completion 2027-12-16 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment-Emergent adverse event (TEAE) and serious adverse event (SAE) | From first dose until last visit(within 85 days after drug injection)
  Adverse event (AE) will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0.The safety profile of LBL-047 will be assessed by monitoring the adverse event (AE) and serious adverse event (SAE) During treatment.

SECONDARY OUTCOMES:
Cmax | From first dose until last visit(within 85 days after drug injection)
  Maximum drug concentration in plasma after administration.
Tmax | From first dose until last visit(within 85 days after drug injection)
  After administration,Time to reach maximum drug concentration in plasma.
Immunogenicity | From first dose until last visit(within 85 days after drug injection)
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects.Immunogenicity refers to the performance that can elicit an immune response.
Assessment of Pharmacodynamics | From first dose until last visit(within 85 days after drug injection)
  Drug therapy effect and adverse reaction, such as B cell level.

CONTACTS AND LOCATIONS:
Overall Officials: xianmin meng, Principal Investigator — Shanghai Public Health Clinical Center
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No